CLINICAL TRIAL: NCT03144180
Title: Compare the Q-Cup With Other Umbilical Cord Blood Collection Techniques: A Feasibility Study
Brief Title: Compare the Q-Cup With Other Umbilical Cord Blood Collection Techniques
Acronym: qcup
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Sireesha Reddy, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E17020
Record Dates: First submitted 2017-05-04; First posted 2017-05-08 (Actual); Results first posted 2020-01-09 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2019-12

CONDITIONS: Pregnant
Keywords: pregnant; third trimester; umbilical cord blood collection

STUDY DESIGN:
Intervention Model Description: Although we tested device feasibility and we should have fewer than 10 participants, we did want to run a two-sided, two-sample t-test with 80% power and an alpha of 0.05, and a common standard deviation of 14 seconds. In order to achieve this, we needed to recruit 30 subjects in total, 15 in the control and 15 in the study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control (No Intervention): The Q-cup will not be used to collect umbilical cord blood.
- Study Group (Active Comparator): The Q-cup will be used to collect umbilical cord blood.
  Interventions: Device: Q-cup

INTERVENTIONS:
Device: Q-cup — This technology is a different way of collecting umbilical cord blood.
  Arms: Study Group

SUMMARY:
Currently there is no standardized method of collecting and transferring umbilical cord blood to laboratory vacuum tubes. Current methods are messy and may require needles to draw the blood presenting risk of blood exposure and percutaneous injury to obstetrical personnel. A safer, more efficient method of collecting cord blood is needed. The investigators propose to use the Q-Cup technology for collecting cord blood. The Q-Cup device is a two-piece injection molded blood collection and transfer device that enables safe and easy collection of blood from the newborn's umbilical cord and readily transfers the blood into a laboratory vacuum tube. The device consists of a collection cup with a wide opening to easily collect blood from the umbilical cord and a guide tube with a recessed needle which is attached to the collection cup. The operator is enabled to fill the required vacuum containing tubes in a clean, quick, efficient and safe manner by simply inserting the vacuum tube into the guide tube of the Q-Cup. As a result, there is less risk of blood exposure and percutaneous injury and blood is collected more efficiently. This device allows the practitioner to collect and transfer umbilical cord blood: without the need for removing the stopper from the vacuum tube (reducing mess and contamination) and without the need for a syringe and exposed needle (reducing injury and infection).

DETAILED DESCRIPTION:
Approximately 4 million babies were born in the United States in 2015. Umbilical cord blood (UBC) collection is a routine hospital procedure done to evaluate a newborn's health after the birth of the fetus. UBC is tested to measure bilirubin levels, blood gases, blood sugar levels, blood types, complete blood counts, and platelet counts. UBC is collected by either draining the blood into the collection vial, milking the umbilical cord of blood, or extracting the blood by injecting a needle with a syringe. The Center for Disease Control (CDC) estimates 5.6 million workers in the health care industry are at risk of occupational exposure to bloodborne pathogens. Occupational exposure during umbilical cord blood collection may occur due to the great deal of blood and amniotic fluid present at the time of delivery. This fluid causes the physician to have a slippery grasp on the umbilical cord and vials for collection. These methods pose a risk of exposing Labor and Delivery staff to blood borne diseases. The drainage and milking method can lead to an increased amount of spilled blood while the extraction method may lead to accidental needle sticks. Exposure to bloodborne pathogens may be amplified when the umbilical cord is engorged with blood and as the needle is inserted in the cord, splatter may occur. The Needlestick Safety and Prevention Act was signed into law on November 6, 2000 in which employees were required to implement safer medical devices. Many patents have been obtained for umbilical cord blood collection devices however, there has not been a standardized method of collecting and transferring umbilical cord blood to the laboratory vacuum tubes. The goal of this project is to prove the feasibility of using the Q-Cup, a patent pending disposable, two-piece blood collection and transfer device for safely and efficiently collecting umbilical cord blood and transferring it into laboratory vacuum tubes.

The overall objective of this project is to prove the feasibility of using a two-piece umbilical blood collection and transfer device for safely and effectively collecting umbilical cord blood and transferring the blood into a laboratory vacuum tube. Also, the investigators will assess provider satisfaction, safety, ease of use, length of procedure comparing passive flow into blood tubes and the Q-cup technology. The Q-Cup technology can take part in the effort to reduce occupation exposures including percutaneous exposures during labor and delivery in general and by studying specifically the heretofore neglected category of umbilical cord blood collection and transfer. Efforts in this area will help focus attention on this previously ignored domain and help establish a standard of care and safety during this frequent procedure.

The investigators hypothesize the Q-Cup will be a more effective transfer method than current practices utilized for umbilical cord blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Obstetric patients must be age 18 or older
* Obstetric patients must be receiving prenatal care at Texas Tech University Health Sciences Center El Paso Department of Ob-Gyn
* Obstetric patients must be in their third trimester
* Obstetric patients must be delivering at University Medical Center

Exclusion Criteria:

* children will not be included
* patients in active labor

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2017-07-19 (Actual); Primary Completion 2017-09-14 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schaffer, MD, Principal Investigator — Texas Tech University Health Sciences Center, El Paso
Locations (1):
- Texas Tech University Health Sciences Center El Paso, El Paso, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Perry J, Jagger J. Collecting umbilical cord blood. Nursing. 2004 Oct;34(10):20. doi: 10.1097/00152193-200410000-00016. No abstract available. PMID 15489606
- [Background] Eder JM, Cutter GR. A new device for collecting cord blood. Obstet Gynecol. 1995 Nov;86(5):850-2. doi: 10.1016/0029-7844(95)00274-U. PMID 7566863
- See also: cord blood — https://medlineplus.gov/ency/article/003403.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at an academic medical center between July 2017 and August 2017. The first participant was enrolled on July 19, 2017 and the last participant was enrolled on August 24, 2017.
Pre-assignment Details: Of the 32 enrolled participants, 16 were randomized to the study arm.
Groups:
- Control: The standard of care methods of umbilical cord collection was used. These include: 1) milking the blood from the umbilical cord into an open specimen tube 2) holding the umbilical cord over a basin and letting blood drip into it, then drawing up the blood into a needless syringe 3) Holding the umbilical cord over a specimen tube and letting the blood drip into it 4) using a conventional needle and syringe to draw blood directly from the cord.
- Study Group: Umbilical cord blood was collected using the Q-cup device.
Period: Overall Study
Arm/Group | Control | Study Group
Started | 16 | 16
Completed | 14 | 10
Not Completed | 2 | 6
Not completed — STAT Delivery | 1 | 1
Not completed — Provider forgot to fill out forms | 1 | 3
Not completed — Provider forgot to use the Q-cup | 0 | 1
Not completed — Scrub tech removed tube cap | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Study Group | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 16 | 16 | 32
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Participants Delivery Provider [Count of Participants; unit: Participants] — A Demographic survey was self-administered by the delivery provider, however, some delivery providers did not fill out the surveys and therefore, data was missing.
  Participants
    Delivered by Faculty | 10 | 6 | 16
    Delivered by Resident | 2 | 4 | 6
    Delivered by Unknown | 4 | 6 | 10
Delivery Type [Count of Participants; unit: Participants] — A Demographic survey was self-administered by the delivery provider, however, some delivery providers did not fill out the surveys and therefore, data was missing.
  Participants
    Vaginal Delivery | 14 | 9 | 23
    Cesarean Section | 0 | 2 | 2
    Missing | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Mean Blood Collection Time
Description: Anticipating the average lengths of cord blood collection with the standard method is 15 seconds and 30 seconds with the Q-cup, we needed 30 subjects total. 15 in the Q-cup arm of the study and 15 in the comparison group (for a two-sided two-sample t-test with 80% power, an alpha of 0.05, and a common standard deviation of 14 seconds). 30 participants were recruited into the study, however, the delivery providers were in charge of collecting this outcome.
Time Frame: 12 weeks
Population: All participants were assigned to the standard of care or the q-cup. The delivery providers collected this outcome.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- Standard of Care (Control): A timer was used to measure how long (in seconds) it took for the collection tube to fill up with umbilical cord blood using the standard methods.
- Q Cup (Study): A timer was used to measure how long (in seconds) it took for the collection tube to fill up with umbilical cord blood using the Q-cup device.
Arm/Group | Standard of Care (Control) | Q Cup (Study)
Number analyzed (Participants) | 14 | 10
Seconds | 49 (47) | 44 (25)
Statistical Analysis 1: Comparison: Q Cup (Study); Test type: Equivalence — A two-sided two-sample t-test with 80% power, an alpha of 0.05, and a common standard deviation of 14 seconds was used to determine the sample size; Confidence Interval for a mean = 49, 95% CI 2-sided [15.459 to 82.571], Standard Deviation 47

2. Secondary Outcome: Determining Umbilical Cord Collection Cleanliness With the Q-cup as Compared to the Standard Blood Collection Method
Description: Participants' delivery providers were asked to self-administer a survey in which they were to assess blood collection for cleanliness. Possible choices were excellent/ good or fair/poor. Some delivery providers did not fill out the surveys and therefore, data was missing.
Time Frame: At Delivery which could be between 1 to 12 weeks after Baseline.
Population: All participants randomized to Standard of Care or Qcup. Delivery Providers filled out the survey in regards to the collection method.
Measure: Count of Participants; unit: Participants
Groups:
- Standard of Care (Control): The Q-cup will not be used to collect umbilical cord blood.
- Q-cup (Study): The Q-cup will be used to collect umbilical cord blood.
  Q-cup: This technology is a different way of collecting umbilical cord blood.
Arm/Group | Standard of Care (Control) | Q-cup (Study)
Number analyzed (Participants) | 14 | 11
Participants
  Excellent/ Good | 7 | 10
  Fair/ Poor | 7 | 1
Statistical Analysis 1: Comparison: Standard of Care (Control) vs Q-cup (Study); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.0295, Chi-squared — The threshold for statistical significance was p = 0.05

3. Secondary Outcome: Fill Capacity of Umbilical Cord Blood Using the Qcup Compared to Standard of Care
Description: Participant delivery providers were asked to self-administer a survey in which they were to assess the fill capacity of the lab tubes using the Qcup or the standard method. Possible choices were filled to capacity and not filled to capacity. Some delivery providers did not fill out the surveys and therefore, data was missing.
Time Frame: 12 weeks
Population: All participants randomized to Standard of Care or Qcup. Delivery Providers filled out the survey in regards to the fill capacity.
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care (Control) | Q-cup (Study)
Number analyzed (Participants) | 14 | 11
Participants
  Tube Filled to Capacity | 11 | 10
  Tube Not Filled to Capacity | 3 | 1
Statistical Analysis 1: Comparison: Standard of Care (Control) vs Q-cup (Study); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.403, Chi-squared — The threshold for statistical significance was p = 0.05

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Groups:
- Standard of Care (Control): Participants were randomized into the standard of care group in which the Qcup was not used to collect umbilical cord blood by the delivery provider.
- Qcup (Study): Participants were randomized into the study group in which the Qcup was used to collect umbilical cord blood by the delivery provider.
Arm/Group | Standard of Care (Control) | Qcup (Study)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Recruiting patients at the clinic, not at hospital; The patient forgot to tell the triage team they were on the study; At times the Participants' delivery providers forgot to fill out the surveys.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-25): https://cdn.clinicaltrials.gov/large-docs/80/NCT03144180/Prot_SAP_000.pdf